CLINICAL TRIAL: NCT00169338
Title: Pallidal Stimulation in Patients With Post-anoxic and Idiopathic Dystonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marie-laure Welter (Other)
Responsible Party: Sponsor-Investigator, Marie-laure Welter, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Organization: Groupe Hospitalier Pitie-Salpetriere (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P020918
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Dystonia
Keywords: Dystonia; deep brain stimulation; globus pallidus; Post-anoxic dystonia
MeSH Terms: conditions — Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- deep brain stimulation (Experimental): Paladin deep brain stimulation
  Interventions: Procedure: Deep brain stimulation
- sham deep brain stimulation (Placebo Comparator): no stimulation

INTERVENTIONS:
Procedure: Deep brain stimulation — internal pallidal deep brain stimulation
  Arms: deep brain stimulation

SUMMARY:
Bilateral pallidal stimulation is effective in the treatment of patients with generalised idiopathic dystonia. The aim of this study is to evaluate the efficacy of bilateral pallidal stimulation in patients with post-anoxic generalised dystonia or non-generalised primary dystonia.

DETAILED DESCRIPTION:
Evaluate the effect of bilateral pallidal stimulation on the motor disability of patients with post-anoxic generalised dystonia or primary dystonia.

ELIGIBILITY:
Inclusion Criteria:

* Post-anoxic generalised dystonia
* Idiopathic non-generalised dystonia
* Disease duration > 1 year

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI)
* Mini-mental status (MMS) < 24
* Severe psychiatric disorder

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Vidailhet, MD, PhD, Study Director — Hôpital Saint-Antoine
Locations (1):
- Centre d'Investigation Clinique-Hôpital Pitié-Salpetriere, Paris, France